CLINICAL TRIAL: NCT01337141
Title: Multicentric Intervention Study Evaluating the Efficiency of the Implementation in the Spanish Health System of a Telematic System Applied to Metabolic Control Optimization for Type 1 Diabetes Mellitus (DM1) Patients
Brief Title: A Telematic Program for Optimization of Metabolic Control in Diabetes Mellitus Type 1 (DM1) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Biomedical Research Centre in Diabetes and Associated Metabolic Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBERDEM-TELEMED-DIABETES
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 1; Metabolic Disorder
Keywords: Telemedicine; Type 1 diabetes; Metabolic control optimisation; Health care costs; Intervention study; Access to internet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional telematic (Experimental): 80 patients will be included in this arm. They will receive 5 telematic visits (Telecare system) and 2 face to face visits.
  Interventions: Device: Telecare system
- Control (Other): 80 patients will be included in this arm. They will receive 7 face-to-face visits (not telematic).
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — 7 face-to-face visits.
  Other Names: Control group do not use telematic system.
  Arms: Control
Device: Telecare system — 5 telematic visits and 2 face-to-face visits.
  Other Names: Medical Guard Diabetes®; - Access in internet: https://www.medicalguard.net/; - Pulso Ediciones SL
  Arms: Interventional telematic

SUMMARY:
A greater visit frequency between the diabetes mellitus 1 (DM1) patient and the medical team increases the possibilities to improve metabolic control. The support of telematic visits can support the patient and the health system.

Patients and Method: 160 patients (from 5 participating centres) with type 1 diabetes mellitus (DM1) candidates for improved metabolic control selected according to inclusion and exclusion criteria. The telecare system used is comprised of the patient Unit and the doctor Unit. The system allows the patient to send glucose values, insulin doses, carbohydrate contribution and other events via the internet. Both the patient and the professional can use this information via the telecare system platform.

Work hypothesis

The application of interactive telematic systems between patient-health team will improve the cost effectiveness of care programmes for optimisation of metabolic control directed towards diabetes mellitus (DM1) patients.

Objectives:

General Objective Evaluate the impact of the telecare system on the efficiency of economic and clinical management of human and material resources directed to a program of metabolic control optimisation in diabetes mellitus 1 (DM1) patients as well as the level of metabolic control and the quality of life of the patients.

Specific objectives

1. To identify and analyse the influence of the telecare system on patient costs in time, money and normal work or school activity which the patient has to stop to carry out the physical visits for following the programme.
2. To identify and analyse the influence of the telecare system on medical team costs in time, money and care organisation directed towards the monitoring phase of the metabolic control care programme.
3. To identify and analyse the influence of the telecare system on the level of metabolic control: Glycosylated haemoglobin and the presence of acute hypoglycemic and hyperglycaemic complications in diabetes mellitus 1 (DM1) patients that follow the metabolic optimisation programme.
4. To identify and analyse the influence of the telecare system on the quality of life of the patient measured in satisfaction scale, impact, social/work concern and concern relating to diabetes.
5. To identify and analyse the influence of the telecare system on the adherence to different treatment components.

DETAILED DESCRIPTION:
*Title: Multicentric random, prospective, open and comparative intervention study evaluating the efficiency of the implementation in the Spanish Health System of a telematic system applied to metabolic control optimization for type 1 diabetes mellitus (DM1) patients.

* Protocol:

  1) Pre-intervention. After the patient is informed and accepts the protocol they make 2 visits for planning individual treatment. 2) Random Assignment in 2 Groups: A) Intervention (telecare system). B) Control. The intervention group patients will be trained in the telecare system machine. Both groups will make the same number of 6 visits over 6 months: Intervention Group (5 telematics and 1 hospital), Control group (6 hospital). Results will be assessed at 3 and 6 months and reassessed at 12 months.
* Patients The objective of the present study is to demonstrate that telematic control of diabetes mellitus is not inferior to the face to face visit control system, while showing an added value an important reduction in costs. Cost information from three studies have been used for the calculation of the sample 2,3,20 in diabetes mellitus 1 (DM1) patients, some followed in a telematic form (210 ± 184€) and other in the form of face to face visits (376 ± 278€). Relating to this, 72 patients per group are needed to obtain a statistical power of 99% and an alpha level of 0.05 (two-sided). 80 patients per group will be needed to be randomised taking into account a 10% loss percentage.

Participating Centres

* Hospital Clínico. Barcelona
* Hospital Clínico. Valencia
* Hospital Carlos Haya. Málaga
* Hospital Clínico. Madrid
* Hospital de Cruces. Barakaldo

Each arm will include 80 patients, 160 as a total.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus 1 (DM1) patients with more than 5 years of evolution with values of glycosylated haemoglobin (HbA1c) > 8% aged between 18 and 50 years.
* Undergoing treatment with multiple doses of insulin.
* Having 3-4 blood sugar tests per day.
* Suitable knowledge about diabetes (test of Diabetes knowledge questionnaire (DKQ2)>25).
* Patients with a computer and access to home internet.

Exclusion Criteria:

* Pregnant diabetes mellitus 1 (DM1) patients.
* History of severe hypoglycemia.
* Manipulation of results.
* Psychiatric disorder.
* Incapable of carrying out intensive therapy monitoring.
* Physical and/or visual incapacity.
* Participating in another study.
* Patients with infertility treatment (ISCI).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Optimise metabolic control | Month 12
  * Insulin dose and criteria (timetables, habits of diet and activity).
  * Autocontrol description and survey about perception of hypoglycaemia
  * Knowledge about diabetes: Diabetes knowledge questionnaire (DKQ2) <25/35

SECONDARY OUTCOMES:
Patient costs | Month 6
  Time, expenses and ordinary activity (studies and work) that the patient could not do in order to attend to the face-to-face visits.
Medical team costs | Month6
  Time, expenses and healthcare issues used in the follow-up phase of the metabolic control.
Quality of life | Month 12
  Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL) and standardised instrument for use as a measure of health outcome (EuroQoL).
Treatment adherence | Month 12
  Self-Care Inventory-revised (SCI-R), a self-report measure of perceived adherence to diabetes self-care recommendations, among adults with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Enric Esmatjes, MD and PhD, Principal Investigator — Hospital Clínic de Barcelona (CIBERDEM)
Locations (5):
- Spain (5):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Clínico de Madrid, Madrid, Madrid
  - Hospital de Cruces, Barakaldo, Spain
  - Hospital Carlos Haya, Málaga, Spain
  - Hospital Clínico de Valencia, Valencia, Spain

REFERENCES:
- See also: CIBERDEM website, including a description of TELEMED-DIABETES — http://www.ciberdem.org